CLINICAL TRIAL: NCT05288712
Title: Effectiveness of a Training Protocol With the Cervical Device in Subjects With Deep Cervical Muscle Strength Deficit in Cervical Range of Motion, Muscle Endurance and Neck Disability.
Brief Title: Effectiveness of a Training Protocol With the Cervical Device in Subjects With Deep Cervical Muscle Strength Deficit.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Pilar Pardos Aguilella, Collaborating Teacher, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C.P. - C.I. PI21/357
Record Dates: First submitted 2022-03-10; First posted 2022-03-21 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2023-08

CONDITIONS: Muscle Weakness; Cervical Disability
Keywords: neck pain; exercise therapy; muscle weakness; telerehabilitation; neck muscles
MeSH Terms: conditions — Muscle Weakness; Neck Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial with 3 different groups
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental: Training protocol with the cervical device for treatment (CDAT). (Experimental): Endurance and stabilization training program of deep cervical flexors with the cervical device for treatment.
  Endurance and stabilization training program of deep cervical extensors with the cervical device for treatment.
  Interventions: Other: Training protocol with the device cervical for treatment (CDAT)
- Conventional training protocol: (Active Comparator): Endurance and stabilization training program of deep cervical flexors with conventional protocol.
  Endurance and stabilization training program of deep cervical extensors with conventional protocol.
  Interventions: Other: Conventional training protocol
- Control Group (No Intervention): Subject continues with activities of daily living. Does not receive deep cervical muscle training.

INTERVENTIONS:
Other: Training protocol with the device cervical for treatment (CDAT) — Training protocol with the cervical device for treatment (CDAT)
  Arms: Experimental: Training protocol with the cervical device for treatment (CDAT).
Other: Conventional training protocol — Conventional training protocol
  Arms: Conventional training protocol:

SUMMARY:
The purpose of this study is to evaluate the clinical results produced by a training protocol with the new device for cervical treatment (CDAT) and the conventional training protocol (CT) versus a control group (C) in subjects with cervical deep muscle strength deficit and mild neck disability.

DETAILED DESCRIPTION:
Cervical pain is in many cases a decrease in the quality of life.The cervical spine is the most mobile region of the spine which also must be strong enough in order to support the weight of the skull. Deficits in deep cervical muscle strength are related to different clinical conditions: cervicogenic dizziness, cervical radiculopathy, cervical mechanical-chronic, cervical pain and cervical instability. Training protocols can help to improve pain, cervical function, posture and cross-sectional area. However, there are no training protocols in subjects with mild disability and strength deficit of the deep cervical muscle, including deep neck extensor and flexor muscles. The cervical device treatment (CDAT) allows us to train the cervical flexor and extensor muscle in a simple and comfortable way.

ELIGIBILITY:
Inclusion Criteria:

* Deep flexor strength deficit in craniocervical flexion test.
* Deep extensor strength deficit in neck extensor muscle endurance test.
* ≤ 14 score in Neck disability Index.

Exclusion Criteria:

* Have received cervical treatment during the last six month, presented any red flag, neurological or cognitive impairment (inability to understand the questionnaires or examination).
* Have received cervical manual therapy treatment during the last six month.
* A history of cervical trauma or surgery during the last year.
* Chronic neck pain occurring during the last six months (intensity, visual analogue scale >3/10, frequency > 2 days/week, duration >3 hours/day).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-09-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | Baseline and 6 weeks, 10 weeks, 14 weeks
  Mean change from baseline in Neck Disability Index (NDI) (Neck Function) after 6 weeks , 10 weeks and 14 weeks.
  The examiners assess the self-perceived disability from neck pain using the NDI. The Neck Disability Index (NDI) is designed to measure neck-specific disability. The questionnaire has 10 items concerning pain and activities of daily living including personal care, lifting, reading, headaches, concentration, work status, driving, sleeping and recreation. The measure is designed to be given to the patient to complete.
  Item scores range from 0 (no disability) to 5 (total disability), with the minimum score is 0 (no disability) and maximum score of 50 (complete disability).
Cervical Spine range of motion | Baseline and 6 weeks, 10 weeks, 14 weeks
  Mean change from baseline in Lower and Upper Cervical Spine Range of Movement (ROM) after 6 weeks , 10 weeks and 14 weeks.
  The examiners assess the cervical ROM using CROM (Cervical Range-of-Motion Instrument). Cervical flexion, extension, right/left sidebending, right/left rotation will be evaluated.
  The examiners assess the cervical ROM using CROM (Cervical Range-of-Motion Instrument). Upper cervical flexion, upper cervical extension and flexion rotation test will be evaluated. Flexion rotation test is used to see the amount of movement of the upper cervical spine and is the test most used in the literature. It is positive when there is a decrease of 10 degrees or more in the cervical rotation with maximum flexion, in a sense with respect to the contralateral or presents hypomobility of segment C1 with a mobility less than 32.
Craniocervical flexion test | Baseline and 6 weeks, 10 weeks, 14 weeks
  The examiners assess the strength of deep cervical flexors with craniocervical flexion test.
GLOBAL RATING OF CHANGE SCALE (GROC) | Baseline and 6 weeks, 10 weeks, 14 weeks
  The examiners assess self-perceived improvement in a patient and has been used as an anchor method to determine minimal clinically important change scores after 6 weeks, 10 weeks and 14 weeks. The GROC is a single-item, recall-based questionnaire of well-being that is based on progress (or lack of progress) since an initial treatment encounter.
  Item scores range from - 7 (A very great deal worse) to + 7 A very great deal better.

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Pardos-Aguilella, teacher, Principal Investigator — UicCatalunya
Locations (1):
- Élite Fisioterapia, María Montessori 2., Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No